CLINICAL TRIAL: NCT06832514
Title: An Investigator-initiated, Single-center Academic Study in Healthy Transgender and Cisgender Persons Aged Between 18 and 50 Years to Investigate Gender and Sex Differences in Immune Responses to Meningococcal Serogroup B Vaccination
Brief Title: Investigating Gender and Sex Differences in Immune Responses Through Vaccination of Transgender and Cisgender Persons
Acronym: Vaxxygender
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University Ghent (Other)
Collaborators: University Hospital, Ghent (Other); Centre for Vaccinology - CEVAC (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: ONZ-2024-0461; 2024-515599-11-00 (EU CTIS Number)
Record Dates: First submitted 2025-02-10; First posted 2025-02-18 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Meningococcal Meningitis, Serogroup B; Transgender Persons; Sex Differences in Immune Response; Vaccination
Keywords: Gender
MeSH Terms: conditions — Meningitis, Meningococcal; Coitus | interventions — 4CMenB vaccine

STUDY DESIGN:
Intervention Model Description: A total of 250 healthy adults will be recruited, with 120 completing the trial, and divided in the following 4 cohorts, each consisting of 30 healthy adult participants aged 18-50 years (inclusive):
  * Cohort 1: Transgender men (n=30)
  * Cohort 2: Transgender women (n=30)
  * Cohort 3: Cisgender men (n=30)
  * Cohort 4: Cisgender women (n=30) Each particpant will receive the four-component meningococcal serogroup B (4CMenB, Bexsero) vaccine as two intramuscular doses, with a one month interval.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- 4CMenB vaccination cisgender men (Experimental): The four component meningococcal serogroup B (4CMenB) vaccine will be administered to 30 cisgender men via two intramuscular injections, with a one month interval.
  Interventions: Biological: Serogroup B meningococal vaccine
- 4CMenB vaccination cisgender women (Experimental): The four component meningococcal serogroup B (4CMenB) vaccine will be administered to 30 cisgender women via two intramuscular injections, with a one month interval.
  Interventions: Biological: Serogroup B meningococal vaccine
- 4CMenB vaccination transgender women (Experimental): The four component meningococcal serogroup B (4CMenB) vaccine will be administered to 30 transgender women via two intramuscular injections, with a one month interval.
  Interventions: Biological: Serogroup B meningococal vaccine
- 4CMenB vaccination transgender men (Experimental): The four component meningococcal serogroup B (4CMenB) vaccine will be administered to 30 transgender men via two intramuscular injections, with a one month interval.
  Interventions: Biological: Serogroup B meningococal vaccine

INTERVENTIONS:
Biological: Serogroup B meningococal vaccine — The 4CMenB vaccine will be administered via two intramuscular (IM) injections in the non-dominant upper arm, with a one month interval.
  Other Names: Four component meningococcal serogroup B vaccine; 4CMenB; Bexsero

SUMMARY:
Sexual differences are a well-established source of biological variation in immune system functioning, with men often displaying lower adaptive immune responses (e.g. antibody production) to infections and vaccinations compared to women. The impact of sex and gender on immune responses and immune functioning warrants more in-depth investigation. This study is an investigator-initiated project aimed at prospectively assessing the immune response towards a vaccine in transgender and cisgender individuals. Transgender individuals retain their chromosomal sex while undergoing a significant hormonal shift that aligns with their experienced gender. Immune responses induced by the four-component meningococcal serogroup B (4CMenB; Bexsero®) vaccine will be evaluated in transgender individuals and compared with responses observed in cisgender individuals. Both humoral and cellular immune responses induced by two doses of the 4CMenB vaccine will be quantified and analysed. This approach is expected to provide new insights into the effects of gender and sex differences on innate and adaptive immune responses.

ELIGIBILITY:
Inclusion Criteria:

1. Written signed informed consent form (ICF) obtained before any study-related activities.
2. Participants aged between, and including, 18 and 50 years of age at the time of signing the ICF which equals with the time of the first study intervention.
3. Participants who are considered to be in good general health as determined by the investigator by medical evaluation including medical history andphysical examination at enrollment.
4. Participants with a BMI within the range 18.5 to 35 kg/m2 inclusive at screening.
5. POCBP (18-50 years of age) who are not pregnant or breastfeeding or planning to become pregnant during the clinical study.
6. Transgender persons need to be under stable gender-affirming hormone therapy (GAHT) for at least 6 months. Compliance needs to be documented by hormonal lab tests.
7. POCBP must have a negative urine pregnancy test at each vaccination visit (Visit 1 and Visit 5) Refer to Section 8.6.5 for Pregnancy Testing.
8. Participants who are willing and able to comply with the study procedures and are capable to comply with the requirements of the protocol (e.g. return for follow-up visits) as determined by the investigator.

Exclusion Criteria:

1. Current or previous, confirmed or suspected disease caused by N. meningitidis and N. gonnorrhoea.
2. Household contact with and/or intimate exposure (e.g. sexual or saliva contact) to an individual with laboratory confirmed N. meningitidis infection during life.
3. Transgender persons in a diagnostic phase (no hormonal intervention) or undergoing treatment based on the suppression of endogenic hormones (e.g. gonadotropin releasing hormone analogues).
4. Current or previous infection with hepatitis B, hepatitis C or human immunodeficiency virus (HIV) as determined by anamnesis and medical history.
5. Past or current confirmed or suspected immune-suppressive or immune-deficient condition, at the discretion of the investigator, including but not limited to blood, endocrine, hepatic, muscular, nervous system or skin autoimmune disorders, lupus erythematosus and associated conditions or disorders (e.g. rheumatoid arthritis, scleroderma) or immunodeficiency syndromes (including, but not limited to: acquired immunodeficiency syndromes and primary immunodeficiency syndromes).
6. History of confirmed hypersensitivity, anaphylaxis and/or other severe allergic reactions (e.g., generalized urticaria, angioedema, bronchospasm) to any component of the study vaccine or excipients (sodium chloride, histidine, sucrose, kanamycin and water for injection), medical products, or medical equipment whose use is foreseen in this study, as determined by the investigator.
7. Clinical conditions representing a contraindication for IM administration and blood draws, as judged by the investigator, e.g. thrombocytopenia or history of bleeding disorder (e.g. factor deficiency, coagulopathy, or platelet disorder requiring special precautions) or significant bruising or bleeding difficulties.
8. History of asplenia, functional asplenia or any condition resulting in the absence or removal of the spleen.
9. Active malignancy or malignancy within the past 5 years that, in the opinion of the investigator, may affect immune response or participant safety - except for localized and fully treated cancers not requiring long-term therapy such as chemotherapy or radiotherapy (e.g. completely resected basal cell carcinoma, cervical intraepithelial neoplasia, melanoma in situ, early-stage thyroid cancer), based on the investigator's clinical judgement.
10. History of idiopathic urticaria within the past year.
11. Currently pregnant, breast-feeding or planning to become pregnant. Cisgender women with permanent infertility due to an alternate medical cause (e.g. documented bilateral oophorectomy, androgen insensitivity, gonadal dysgenesis) are excluded to participate. For individuals with permanent infertility due to an alternate medical cause other than the above, investigator discretion should be applied to determining study entry. Additionally, cisgender women in a postmenopausal state, defined as no menses for 12 months without an alternative medical cause are also excluded to participate. Refer to
12. Any other clinical condition that, in the opinion of the investigator, could compromise the participant's safety and/or compliance with the study protocol (e.g. current or recent (< 1 years ago) heavy smoking (> 20 cigarettes per day) or daily heavy vaping (equivalent to 20 cigarettes), drug- or alcohol (> 15 units for cisgender men and transgender women or > 10 units or cisgender women and transgender men per week) abuse/addiction.
13. Behavioral or cognitive impairment, unstable psychiatric conditions (e.g. forced admission, suicidal thoughts in the last two year) or other psychiatric disease that, in the opinion of the investigator, may interfere with study compliance, as well as with the subject's ability and/or safety to participate in the study. Stable psychiatric conditions (e.g. under-controlled depression) will be evaluated based on the investigators judgement.
14. Donation of blood or blood products within 90 days prior to the first vaccination visit (Visit 1) until Day 56 (Visit 9).
15. Previous vaccination against any group B meningococcal vaccine (Bexsero®, Trumenba®) at any time prior to informed consent.
16. Prior receipt of a live-attenuated vaccine in the 28 days prior to administration of the 4CMenB vaccine, within 14 days for subunit or inactivated vaccines or planning to receive a vaccine in between the first and second vaccine administration, as well as 28 days following administration of the second 4CMenB vaccine dose.
17. Currently participating in another clinical study, or planning to participate in another study during the study period, or administration of any investigational drug or medical device in the 28 days prior to study vaccination.
18. Prior receipt of blood, blood-derived products or immunoglobulins in the 6 months prior to administration of the study vaccine, or planning to receive such product during the study period.
19. Chronic administration (defined as 14 consecutive days in total) of immunosuppressants (e.g. corticosteroids (PO/IV/IM) or other immune-modifying drugs (e.g. antineoplastic agents, radiotherapy) during the period starting 90 days prior to vaccination or planned administration during the study (excluding topical, inhaled and intranasal preparations and intra-articular injections). For corticosteroids, this will mean prednisone ≥ 20 mg/day, or equivalent.
20. POCBP (cisgender women and transgender men) who use the following contraceptive methods will not be included in the study

    * Oral, injectable, intravaginal (i.e. intravaginal ring) or transdermal combined (oestrogen- and progesterone-containing) hormonal contraception associated with inhibition of ovulation.
    * Oral, injectable or implantable progestogen-only hormonal contraception associated with inhibition of ovulation.
21. Current anti-tuberculosis prophylaxis or therapy.

25. Participants with a history of any medical conditions that, in the opinion of the investigator, might interfere with the results of the study or pose additional risk to the participants when participating in the study.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 250 (Estimated)
Dates: Start 2025-01-31 (Actual); Primary Completion 2026-07-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Characterise humoral, adaptive immune responses elicited by two administrations of 4CMenB in transgender and cisgender healthy participants, aged 18 to 50 years. | From the first vaccination visit to two months post-primary vaccination
  The human serum bactericidal antibody titers (hSBA) against reference strains for factor H binding protein (fHbp), Neisseria adhesin A (NadA) and Porine A (PorA) in transgender and cisgender participants.

SECONDARY OUTCOMES:
Characterise the cellular (CD4+ and CD8+ T cell), adaptive immune responses elicited by two administrations of 4CMenB in transgender and cisgender healthy participants, aged 18 to 50 years. | From the first vaccination visit to two months post-primary vaccination
  T cell-mediated immune responses in peripheral blood mononuclear cells (PBMCs) collected at different timepoints post-vaccination in 4CMen-B vaccinated transgender and cisgender participants.

OTHER OUTCOMES:
Characterise innate immune responses elicited by two administrations of 4CMenB in transgender and cisgender healthy participants, aged 18 to 50 years | From the first vaccination visit to seven days post-secondary vaccination
  * White blood cell counts and C-reactive protein levels at Day 0 and 28 (prior to primary and secondary vaccination, respectively), and 1, 3 and 7 days post-primary and secondary vaccination, as well as 56 days post-primary vaccination with 4CMenB in transgender and cisgender participants
  * Cytokine production measured at Day 0 and 28 (prior to primary and secondary vaccination, respectively), as well as 1, 3 and 7 days post-primary and secondary vaccination with 4CMenB between transgender and cisgender participants.
Cellular (CD4+ and CD8+ T cell), adaptive immune responses elicited by two administrations of 4CMenB in transgender and cisgender healthy participants, aged 18 to 50 years. | From 7 days post-primary vaccination to 180 days post-primary vaccination
  T cell-mediated immune responses in PBMCs collected at Day 28 (prior to secondary vaccination), 7 days post-primary and secondary vaccination, as well as 180 days post-primary vaccination with 4CMenB in transgender and cisgender participants as confirmed by the presence of 4CMenB-specific CD4+ and CD8+ T cells producing at least CD40L, IFN-γ, IL-2, and/or TNF-α as measured by flow cytometry (intracellular cytokine staining).
Cellular, regulatory T (Treg) cell immune responses elicited by two administrations of 4CMenB in transgender and cisgender healthy participants, aged 18 to 50 years. | From the first vaccination visit to 180 days post-primary vaccination
  Treg cell-mediated immune responses in PBMCs collected at Day 0 and 28 (prior to primary and secondary vaccination, respectively), 7 days post-primary and secondary vaccination, as well as 56 and 180 days post-primary vaccination with 4CMenB in transgender and cisgender participants, measured by flow cytometry (intracellular cytokine staining).
Changes in gene expression and epigenetic modifications at the single-cell immunological level after administration of 4CMenB in transgender and cisgender healthy participants, aged 18 to 50 years. | From vaccination to 7 days post-primary and secondary vaccination
  Characterization of innate and adaptive immune responses by examining differentially expressed immune genes in PBMCs collected at Day 0 and 28 (prior to primary and secondary vaccination, respectively), 1, 3 and 7 days post-primary and secondary vaccination with 4CMenB in transgender and cisgender participants.
  Characterization of immune responses by examining expressed genes, changes in gene expression levels, changes in epigenetic responses, and enriched/activated pathways in PBMCs collected at Day 0 and 28 (prior to primary and secondary vaccination, respectively), 1, 3 and 7 days post-primary and secondary vaccination with 4CMenB in transgender and cisgender participants.
Characterise local and systemic AEs, SAEs, pIMDs and SUSARs to two administrations of 4CMenB in transgender and cisgender healthy participants, aged 18 to 50 years. | From the first vaccination visit to 180 days post-primary vaccination
  * Occurrence of solicited local and systemic adverse events (AEs), starting from the date of vaccination and the six following days, in all participants (trans- and cis-gender participants).
  * Occurrence of unsolicited AEs, starting from the date of vaccination and the six following days in all participants (trans- and cis-gender participants).
  * Occurrence of serious adverse events (SAEs), potential immune mediated disease (pIMD) and suspected unexpected serious adverse reaction (SUSAR) during the entire study period, i.e. until 180 days (±14 days) post-primary vaccination in all participants (trans- and cis-gender participants).

CONTACTS AND LOCATIONS:
Overall Officials: Prof. Dr. Isabel Leroux-Roels, PhD, MD, Principal Investigator — CEVAC, University Hospital Ghent, Belgium
Locations (1):
- CEVAC, University Hospital Ghent, Belgium, Ghent, Belgium

IPD SHARING:
Plan to Share IPD: No